CLINICAL TRIAL: NCT04381637
Title: Newborn Infant Parasympathetic Evaluation (NIPE) Index After Three Standardized Tetanic Stimulations (10, 30 and 60 Miliamps) Performed in a Randomized Sequence Under General Anesthesia in a Pediatric Population
Brief Title: Newborn Infant Parasympathetic Evaluation (NIPE) Index After Standardized Tetanic Stimulations Under General Anesthesia
Acronym: NIPESTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019_32; 2020-A00295-34 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia
Keywords: Monitoring; General anesthesia; Analgesia; Pain; Pediatric
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Intervention Model Description: The research does not involve the evaluation or comparison of medical strategies.The order of application of the stimuli will be randomized according to a Latin square of order 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIPE (Experimental)
  Interventions: Device: NIPE monitor; Procedure: Tetanic stimulations

INTERVENTIONS:
Device: NIPE monitor — NIPE monitor connected to the anesthetic station. No part of the device in contact with the patient. No action on patient or anesthesia. Automatic recording of Heart rate and NIPE index during the study period.
Procedure: Tetanic stimulations — Three tetanic stimulations will be performed (10-30 and 60 milliamps) under general anesthesia, before surgical incision.
  Stims performed via the muscle relaxation monitor (used in standard practice in this population) Each stim lasts for 5 seconds. Interval between two stims : 3-5 minutes Order on intensities randomized by a latin square of order 3.

SUMMARY:
NIPE monitor is the recently developed pediatric version of the ANI monitor, which is used in adults to monitor analgesia during general anesthesia. In adults, under general anesthesia, ANI decreases after a nociceptive stimulation. The amplitude of this decrease is related to the intensity of the stim. This study aims to investigate if NIPE index decreases in the same manner after stimulations in anesthetized children.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery under general anesthesia requiring tracheal intubation and muscle relaxation
* Written informed consent obtained from parents (and from child if appropriate)

Exclusion Criteria:

* Thoracic or cardiac surgery
* Cardiac arrhythmia, Pace maker
* Analgesic medication less than 24 hours before surgery
* Chronic anticholinergic medication
* Contraindication to muscle relaxants or general anesthetics

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Variation of NIPE index (∆NIPE) | 3 minutes following tetanic stimulation
  ∆NIPE = [NIPE minimal value in the 3 minutes following the stim] - [NIPE before stim]
  NIPE varies from 0 to 100. Monitor displays one value per second. NIPE index expected to decrease after stim.

SECONDARY OUTCOMES:
Heart rate Variation (∆HR) | 3 minutes following tetanic stimulation
  ∆HR = [HR maximal value in the 3 minutes following the stim] - [HR before stim] Heart rate expected to increase after stim.

CONTACTS AND LOCATIONS:
Overall Officials: Anne LAFFARGUE, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France

REFERENCES:
- [Derived] Lebrun S, Boccara J, Cailliau E, Herbet M, Tavernier B, Constant I, Sabourdin N. Quantitative assessment of a pediatric nociception monitor in children under sevoflurane anesthesia. Reg Anesth Pain Med. 2022 Jun 2:rapm-2022-103547. doi: 10.1136/rapm-2022-103547. Online ahead of print. PMID 35654480